CLINICAL TRIAL: NCT00002291
Title: A Double-Blind Group Comparative Study To Evaluate the Safety and Effectiveness of Three Different Doses of Aerosol Pentamidine in the Prophylaxis of Pneumocystis Carinii Pneumonia in Patients With AIDS Post First Episode PCP
Brief Title: The Safety and Effectiveness of Pentamidine in the Prevention of Pneumocystis Carinii Pneumonia (PCP) in Patients With AIDS Who Have Had PCP Before
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisons (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 022A; 87-71
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Dose-Response Relationship, Drug; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To evaluate and compare the safety, tolerability, and efficacy of biweekly administration of 1 of 3 doses of aerosol pentamidine when used as a prophylactic agent in patients who have recovered from their first episode of AIDS-associated Pneumocystis carinii pneumonia (PCP).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at time of entry or those with either of the following AIDS-defining O.I.'s prior to entry:
* Toxoplasmosis.
* Cryptococcosis.
* Transfusion dependent (requiring blood transfusion more than once per month). The last transfusion cannot have been given within 7 days of study entry.
* Pulmonary Kaposi's sarcoma (KS).
* Asthma requiring medication.
* Active therapy for tuberculosis.

Concurrent Medication:

Excluded:

* Active therapy for tuberculosis.

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at time of entry or those with either of the following AIDS-defining O.I.'s prior to entry:
* Toxoplasmosis.
* Cryptococcosis.
* Transfusion dependent (requiring blood transfusion more than once per month). The last transfusion cannot have been given within 7 days of study entry.
* Pulmonary Kaposi's sarcoma (KS).
* Unwilling to sign informed consent.
* Cannot cooperate with study procedures.
* Asthma requiring medication.

Prior Medication:

Excluded within 30 days of study entry:

* Antiretrovirals other than zidovudine (AZT).
* Immunomodulating agents.
* Corticosteroids.

Patients must:

* Have AIDS and recovered from their first episode of cytologically or histologically proven Pneumocystis carinii pneumonia (PCP).
* Be at least 2 weeks and no more than 24 weeks status post therapy for acute PCP.
* Have positive antibody to HIV by any federally licensed ELISA test kit, or confirmed Western blot test.
* Have adequate pulmonary function (vital capacity = or > 80 percent of predicted; forced expiratory volume (FEV), 1 s = or > 65 percent of total FEV; and corrected pulmonary diffusion capacity > 60 percent of predicted).
* Free of acute medical problems.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Fisons Corp, Rochester, New York, United States

REFERENCES:
- [Background] Murphy RL, Lavelle JP, Allan JD, Gordin FM, Dupliss R, Boswell SL, Waskin HA, Davies SF, Graziano FM, Saag MS, et al. Aerosol pentamidine prophylaxis following Pneumocystis carinii pneumonia in AIDS patients: results of a blinded dose-comparison study using an ultrasonic nebulizer. Am J Med. 1991 Apr;90(4):418-26. PMID 2012082